CLINICAL TRIAL: NCT02048358
Title: Randomized, Double-blind, Placebo- and Active Comparator- Controlled Crossover Study in Healthy Male Subjects and an Open Label Study in Healthy Subjects and MS Patients to Assess the Safety, Pharmacokinetics and Pharmacodynamics of 2B3-201
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics Study With 2B3-201 in Healthy Subjects and Multiple Sclerosis(MS) Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: BBB-Therapeutics B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2B3-201-CR-001; 2013-004077-28 (EudraCT Number)
Record Dates: First submitted 2014-01-17; First posted 2014-01-29 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Volunteers; Multiple Sclerosis
Keywords: Healthy volunteers; first in human; 2B3-201; methylprednisolone; CNS-targeting; liposomal; crossover; placebo controlled; active controlled; multiple sclerosis; multiple sclerosis relapse
MeSH Terms: conditions — Multiple Sclerosis | interventions — Glucose; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- 2B3-201 150mg (Experimental): 2B3-201 150mg, once, IV infusion in 1000ml 5% dextrose/ Methylprednisolone hemisuccinate 1000mg, once, IV infusion in 1000ml 5% dextrose/ Placebo, once, IV infusion 1000ml 5% dextrose
  Interventions: Drug: 2B3-201; Drug: Placebo; Drug: Methylprednisolone hemisuccinate
- 2B3-201 300mg (Experimental): 2B3-201 300mg, once, IV infusion in 1500ml 5% dextrose/ Methylprednisolone hemisuccinate 300mg, once, IV infusion in 1500ml 5% dextrose/ Placebo, once, IV infusion 1500ml 5% dextrose
  Interventions: Drug: 2B3-201; Drug: Placebo; Drug: Methylprednisolone hemisuccinate
- 2B3-201 450mg (Experimental): 2B3-201 450mg, once, IV infusion in 2500ml 5% dextrose/ Methylprednisolone hemisuccinate 1000mg, once, IV infusion in 2500ml 5% dextrose/ Placebo, once, IV infusion 2500ml 5% dextrose
  Interventions: Drug: 2B3-201; Drug: Placebo; Drug: Methylprednisolone hemisuccinate
- 450mg 2B3-201 (Experimental): 2B3-201 450mg, once, IV infusion in 2500ml 5% dextrose
  Interventions: Drug: 2B3-201
- 300mg 2B3-201 (Experimental): 2B3-201 300mg, once, IV infusion in 1500ml 5% dextrose
  Interventions: Drug: 2B3-201
- 2B3-201 450mg male volunteers (Experimental): 2B3-201 450mg, once, IV infusion in 1500ml 5% dextrose
  Interventions: Drug: 2B3-201
- 2B3-201 300mg or 450mg female volunteers (Experimental): 2B3-201 300mg or 450mg, once, IV infusion in 1500 or 2500ml 5% dextrose/ Methylprednisolone hemisuccinate 1000mg, once, IV infusion in 1500 or 2500ml 5% dextrose
  Interventions: Drug: 2B3-201; Drug: Methylprednisolone hemisuccinate
- Relapsing MS patients; 2B3-201 450 mg (Experimental): 2B3-201 450mg, once, IV infusion in 2500ml 5% dextrose
  Interventions: Drug: 2B3-201
- Relapsing MS patients; 2B3-201 dose tbd (Experimental): 2B3-201 (dose to be determined), once, IV infusion in 5% dextrose
  Interventions: Drug: 2B3-201

INTERVENTIONS:
Drug: 2B3-201
  Other Names: 2B3-201: glutathione PEGylated-liposomal methylprednisolone
Drug: Placebo
  Other Names: 5% Dextrose
  Arms: 2B3-201 150mg; 2B3-201 300mg; 2B3-201 450mg
Drug: Methylprednisolone hemisuccinate
  Other Names: Solu-Medrol
  Arms: 2B3-201 150mg; 2B3-201 300mg; 2B3-201 300mg or 450mg female volunteers; 2B3-201 450mg

SUMMARY:
In this first in human study the aim is to assess the safety, pharmacokinetics and pharmacodynamics of 2B3-201 in a randomized, first in human, double-blind, placebo- and active comparator- controlled 3-way crossover study in 18 healthy male subjects (part 1). Furthermore, the findings obtained from part 1 will be extended and confirmed in a subsequent parallel open label study in 18 healthy male and 12 MS patients and an open label study with methylprednisolone as comparator in 12 female volunteers (part 2).

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects

* Healthy male or female subjects, 18 to 45 years of age, inclusive. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, and urinalysis.
* Body mass index (BMI) between 18 and 30 kg/m2, inclusive, and with a minimum weight of 50 kg.
* Able to participate and willing to give written informed consent and to comply with the study restrictions.

Relapsing MS patients

* Age: 18 to 65 years, both men and women.
* Patients with relapsing multiple sclerosis (RMS), defined as below, with an acute exacerbation, who in the opinion of the treating physician should undergo a 3 - 5 day course of high dose methylprednisolone;

  * Patients with Relapsing Remitting Multiple Sclerosis (RRMS).
  * Patients with Secondary Progressive Multiple Sclerosis (SPMS) and
  * Patients with clinically isolated syndromes (CIS) who show dissemination of lesions in time (DIT) and space (DIS) on MRI scans according to the 2010 McDonald criteria.
* Able to participate and willing to comply with the study restrictions. Understands and signs the written informed consent prior to any of the testing under this protocol, including screening tests and evaluations that are not considered part of the subject's routine care.

Exclusion Criteria:

Healthy volunteers:

* Any subject who is pregnant or breastfeeding. A urine pregnancy test should be performed in female subjects of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) prior to the start of the study treatment.
* For female subjects of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) and male subjects who are not surgically sterile or with female partners of childbearing potential: absence of effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal gel) will be a contraindication.
* Not willing to use double-barrier contraception, for the duration of the study and for 3 months after the last dose.
* Positive test for drugs of abuse at screening or pre-dose.
* History of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol) within 3 months of screening. Alcohol consumption will be prohibited during study confinement and at least 48 hours before screening, before dosing, and before each scheduled visit.
* History or symptoms of any significant disease including (but not limited to), neurological, psychiatric, endocrine, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder.
* Positive Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening.
* Systolic blood pressure (SBP) greater than 140 mm Hg or less than 90 mm Hg, and diastolic blood pressure (DBP) greater than 90 mm Hg or less than 50 mm Hg.
* Use of any medications (prescription or over-the-counter [OTC]), vitamin, mineral, herbal, and dietary supplements within 21 days of study drug administration. Exceptions are paracetamol (up to 4 g/day).
* Use of CYP3A4-inhibiting drugs, including quinine containing drinks (bitter lemon and tonic water) is prohibited within 21 days of study drug administration
* Subject has used grapefruit, grapefruit juice, grapefruit-containing products, Seville oranges, or pomelo-containing products, within 14 days prior to day -1.
* Clinically significant abnormalities, as judged by the investigator, in laboratory test results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis). In the case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility or judged to be clinically irrelevant for healthy subjects.
* Participation in an investigational drug or device study within 3 months prior to screening.
* Donation of blood over 500 mL within three months prior to screening.
* Concomitant disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study.
* Smoker of more than 10 cigarettes per day prior to screening or who use tobacco products equivalent to more than 10 cigarettes per day.
* Clinically significant abnormal ECG, as judged by the Investigator.
* Current infection or inflammation study within 1 month prior to screening
* Recent vaccinations study within 3 months prior to screening.
* Positive Mantoux test of 5 mm or more.
* Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug, or multiple drug allergies (non-active hay fever is acceptable).
* Unwillingness or inability to comply with the study protocol for any other reason.

RMS patients:

* Previous acute exacerbations, and/or corticosteroid treatment or ACTH < 1 month before present exacerbation,
* Hypersensitivity to methylprednisolone.
* Prior use of immunosuppressive treatments / disease-modifying drugs (DMDs) other than interferon-beta, glatiramer acetate, fingolimod, dimethylfumarate or teriflunomide within 12 months of the index episode. Shorter periods may be allowed at the discretion of the PI and after approval from the sponsor. Subjects may continue their current therapy with interferons, glatiramer acetate, fingolimod, or teriflunomide throughout the course of the study.
* Non-steroidal anti-inflammatory agents, including salicylic acid, should be avoided during the administration of the steroid therapy. If absolutely necessary they are permitted for subjects to treat interferon side effects, when the patient is not responding to acetaminophen/paracetamol.
* Current or recent (within 30 days of first study treatment) treatment with any other investigational drug or participation in any other investigational study
* Evidence of psychiatric illness
* History of any significant cardiac, gastrointestinal, hepatic, pulmonary, renal or active immunosuppressive disease.
* Immune deficiency or any other medical conditions that would preclude corticosteroid therapy.
* Any patient who is pregnant or breastfeeding. A urine pregnancy test should be performed in female subjects of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) prior to the start of the study treatment.
* For female subjects of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) and male subjects who are not surgically sterile or with female partners of childbearing potential: absence of effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal gel) will be a contraindication.
* Physical examination results or laboratory findings that may interfere with the planned treatment, affect patient compliance or place the patient at a high risk of treatment-related complications.
* Known hypersensitivity to any of the cyclodextrin or any excipients in 2B3-201 (e.g. PEG, Cholesterol, HSPC or GSH).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability of 2B3-201 | 3 weeks
  Safety and tolerability of 2B3-201, in comparison to free methylprednisolone hemisuccinate and placebo and the safety and tolerability of 2B3-201amongst the different study populations: healthy male and female subjects and MS patients, additionally the safety and tolerability of 2B3-201 with hydroxypropyl β-cyclodextrin added to the infusion bag will be assessed in healthy male subjects
Pharmacokinetics in plasma of intravenously administered 2B3-201 in terms of Cmax, Volume of distribution, half-life (T1/2), area under the plasma concentration-time curve (AUC), Clearance (CL) | 3 weeks
  Pharmacokinetics of 2B3-201, in comparison to free methylprednisolone hemisuccinate and placebo and the pharmacokinetics of 2B3-201amongst the different study populations: healthy male and female subjects and MS patients. Additionally the pharmacokinetics of 2B3-201 with hydroxypropyl β-cyclodextrin added to the infusion bag will be assessed in healthy male subjects

SECONDARY OUTCOMES:
Measure changes in central nervous system (CNS) functioning after intravenous administration of 2B3-201 by using the Neurocart test battery | 3 weeks
  Neurocart test battery (Pharmaco-EEG, Maze learning, Visual verbal Learning test, Stroop test, Adaptive tracking, VAS Bond & Lader and VAS Bowdle, Eye movements, LSEQ sleep questionnaire) as a measure of pharmacodynamic effects of 2B3-201 on CNS functioning in comparison to free methylprednisolone hemisuccinate and placebo;
Changes in levels of Hypothalamic-pituitary-adrenal (HPA) axis hormones as a measure of pharmacodynamic effects of 2B3-201 in comparison to free methylprednisolone hemisuccinate and placebo; | 3 weeks
Changes in levels of fasting blood glucose as a measure of pharmacodynamic effects of 2B3-201 in comparison to free methylprednisolone hemisuccinate and placebo; | 3 weeks
Changes in levels of osteocalcin concentrations as a measure of pharmacodynamic effects of 2B3-201 in comparison to free methylprednisolone hemisuccinate and placebo; | 3 weeks
Changes in levels of lymphocyte count as a measure of pharmacodynamic effects of 2B3-201 in comparison to free methylprednisolone hemisuccinate and placebo; | 3 weeks
Changes in levels of complement factors during infusion as a measure of pharmacodynamic effects of 2B3-201 in comparison to free methylprednisolone hemisuccinate and placebo; | 3 weeks

OTHER OUTCOMES:
Optimization of the infusion schedule for 2B3-201 with or without the addition of an anti-histaminic drug to minimize the likelihood of non-allergic infusion reactions. | 3 weeks
Changes in neurological examination, Expanded Disability Systems Score (EDSS) and Multiple Sclerosis functional composite (MSFC) after a single dose of 2B3-201 in RMS patients having an acute disease exacerbation, as a measure of clinical efficacy | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Geert-Jan Groeneveld, MD, PhD, Principal Investigator — Center for Human Drug Research
Locations (2):
- Netherlands (2):
  - VUmc, PET and neurology clinical research unit, Amsterdam, North Holland
  - Centre for Human Drug Research (CHDR), Leiden

REFERENCES:
- [Background] Gaillard PJ, Appeldoorn CC, Rip J, Dorland R, van der Pol SM, Kooij G, de Vries HE, Reijerkerk A. Enhanced brain delivery of liposomal methylprednisolone improved therapeutic efficacy in a model of neuroinflammation. J Control Release. 2012 Dec 28;164(3):364-9. doi: 10.1016/j.jconrel.2012.06.022. Epub 2012 Jun 23. PMID 22732475